CLINICAL TRIAL: NCT03079674
Title: China Registry of Non-disabling Ischemic Cerebrovascular Events: A Prospective Multi-center, National Registry Trail
Brief Title: China Registry of Non-disabling Ischemic Cerebrovascular Events
Acronym: CR-NICE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: National Health and Family Planning Commission, P.R.China (Other Government); Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming-Xu, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: GN-2016R0009
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Transient Ischemic Attack; Minor Stroke
Keywords: transient Ischemic Attack; minor Stroke; non-disabling ischemic cerebrovascular events; biomarker; epidemiology; prognosis
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — The faecal samples, plasma, serum and whole blood are retained to establish the biological samples library of NICE.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NICE patients: Non-disabling ischemic cerebrovascular events patients indicate patients with transient ischemic attack and minor stroke (National Institute of Health stroke scale, NIHSS≤3).
  Interventions: Other: observational only- no intervention

INTERVENTIONS:
Other: observational only- no intervention — observational only- no intervention

SUMMARY:
The burden of non-disabling ischemic cerebrovascular events (NICE) is significantly increased. In order to achieve accurate risk stratification and effective treatments, developing new diagnostic, therapeutic, and prognostic strategies is indispensable. Chinese registry of NICE is a national multi-center prospective study aimed to explore the epidemiology, new biomarkers, risk factors and prognostic models.

DETAILED DESCRIPTION:
The pathophysiology of transient ischemic attack (TIA) and minor stroke is a continuous progression. TIA and minor stroke exhibit the common substantial risk factors for early stroke recurrence and epidemiological characteristic. Since TIA and minor stroke may leave impermanent or mild neurological deficit, they are termed as non-disabling ischemic cerebrovascular disease (NICE).

The results of the China Chronic Disease and Risk Factor Surveillance (CCDRFS) 2010 showed that the age-standardized prevalence of TIA is 2.27%. Estimated 23.9 million people may have experienced a TIA in China. The TIA knowing-rate is approximately 3.08% in Chinese adults, only 5.02% received treatment and 4.07% received guideline recommended therapy. The Second China National Stroke Registry (CNSR-II) indicated that minor stroke accounted for 42.23% of all the hospitalized patients of ischemic stroke, which is much higher than that showed in CNSR-I (2007-2008). Thus, it is imperative to develop new strategies to improve the diagnosis, risk prediction and appropriate management of NICE.

NICE is an attractive researching area globally. According to the large quantities of NICE patients in China and the low standardized therapeutic rate, the awareness of NICE is largely insufficient. The purpose of the present study is to establish a multi-center national prospective database of NICE, including clinical information and biological samples library and, to further explore the epidemiology, new biomarkers, risk factors, and prognostic models.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. elapsed time from last episode to registry <48 hours

Exclusion Criteria:

1. patients who refused to participate in the research, and patients who failed to complete the follow-up protocol.
2. patients with malignant tumors, or patients with severe liver or kidney disease, whose life expectancy is less than 1 year.
3. patients who received endovascular or thrombolytic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients (≥18 years) within 48 hours of onset of a minor stroke (National Institute of Health stroke scale, NIHSS≥3) and TIA.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Death | 3 months
  Death from any cause
Death | 6 months
  Death from any cause
Death | 12 months
  Death from any cause
Stroke recurrence | 3 months
  Ischemic stroke
Stroke recurrence | 6 months
  Ischemic stroke
Stroke recurrence | 12 months
  Ischemic stroke

SECONDARY OUTCOMES:
Hemorrhagic stroke | 3 months
  Cerebral hemorrhage and subaraclmoid hemorrhage
Hemorrhagic stroke | 6 months
  Cerebral hemorrhage and subaraclmoid hemorrhage
Hemorrhagic stroke | 12 months
  Cerebral hemorrhage and subaraclmoid hemorrhage
Cardiovascular disease | 3 months
  Coronary heart disease and Angina pectoris
Cardiovascular disease | 6 months
  Coronary heart disease and Angina pectoris
Cardiovascular disease | 12 months
  Coronary heart disease and Angina pectoris
Functional outcome | 3 months
  Modified Rankin Scale ≥3
Functional outcome | 6 months
  Modified Rankin Scale ≥3
Functional outcome | 12 months
  Modified Rankin Scale ≥3

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Xu, MD, PhD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Yilong Wang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (44):
- China (44):
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Shijiazhuang the Third Hospital, Shijiazhuang, Hebei
  - Xingtai Third Hospital, Xingtai, Hebei
  - Anyang People's Hospital, Anyang, Henan
  - The People's Hospital of Hebi, Hebi, Henan
  - The Second People 's Hospital of Jiaozuo, Jiaozuo, Henan
  - The Huaihe Hospital of Henan University, Kaifeng, Henan
  - Luohe Central Hospital, Luohe, Henan
  - Luoyang Central Hospital Affiliated to Zhengzhou University, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang City Central Hospital, Nanyang, Henan
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - The First People's Hospital of Pingdingshan, Pingdingshan, Henan
  - People's Hospital of Puyang, Puyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - The First People's Hospital of Shangqiu, Shangqiu, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Xinyang Central Hospital, Xinyang, Henan
  - Xuchang Central Hospital, Xuchang, Henan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Medical Group of Zhengzhou First People's Hospital, Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Jingmen No.1 People 's Hospital, Jingmen, Hubei
  - Wuhan NO.1 Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - Ankang HospitaL of Traditional Chinese Medicine, Ankang, Shanxi
  - Fenyang Hospital, Fenyang, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Shanxi Provincial People 's Hospital, Xi'an Shi, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - The Institute of Traditional Chinese Medicine of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Yan'an Affiliated Hospital to Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yaghi S, Rostanski SK, Boehme AK, Martin-Schild S, Samai A, Silver B, Blum CA, Jayaraman MV, Siket MS, Khan M, Furie KL, Elkind MS, Marshall RS, Willey JZ. Imaging Parameters and Recurrent Cerebrovascular Events in Patients With Minor Stroke or Transient Ischemic Attack. JAMA Neurol. 2016 May 1;73(5):572-8. doi: 10.1001/jamaneurol.2015.4906. PMID 26998948
- [Background] Meng X, Wang Y, Liu L, Pu Y, Zhao X, Wang C, Wang Y. Validation of the ABCD(2)-I score to predict stroke risk after transient ischemic attack. Neurol Res. 2011 Jun;33(5):482-6. doi: 10.1179/016164111X13007856084043. PMID 21669116
- [Background] Giles MF, Rothwell PM. Risk of stroke early after transient ischaemic attack: a systematic review and meta-analysis. Lancet Neurol. 2007 Dec;6(12):1063-72. doi: 10.1016/S1474-4422(07)70274-0. Epub 2007 Nov 13. PMID 17993293
- [Background] Wu CM, McLaughlin K, Lorenzetti DL, Hill MD, Manns BJ, Ghali WA. Early risk of stroke after transient ischemic attack: a systematic review and meta-analysis. Arch Intern Med. 2007 Dec 10;167(22):2417-22. doi: 10.1001/archinte.167.22.2417. PMID 18071162
- [Background] Wang Y, Zhao X, Jiang Y, Li H, Wang L, Johnston SC, Liu L, Wong KS, Wang C, Pan Y, Jing J, Xu J, Meng X, Zhang M, Li Y, Zhou Y, Zhao W, Wang Y. Prevalence, knowledge, and treatment of transient ischemic attacks in China. Neurology. 2015 Jun 9;84(23):2354-61. doi: 10.1212/WNL.0000000000001665. Epub 2015 May 8. PMID 25957333
- [Background] Wang Y, Cui L, Ji X, Dong Q, Zeng J, Wang Y, Zhou Y, Zhao X, Wang C, Liu L, Nguyen-Huynh MN, Claiborne Johnston S, Wong L, Li H; China National Stroke Registry Investigators. The China National Stroke Registry for patients with acute cerebrovascular events: design, rationale, and baseline patient characteristics. Int J Stroke. 2011 Aug;6(4):355-61. doi: 10.1111/j.1747-4949.2011.00584.x. Epub 2011 Feb 17. PMID 21609414
- [Background] Wang Y, Li Z, Xian Y, Zhao X, Li H, Shen H, Wang C, Liu L, Wang C, Pan Y, Wang D, Prvu Bettger J, Fonarow GC, Schwamm LH, Smith SC Jr, Peterson ED, Wang Y; GOLDEN BRIDGE-AIS investigators. Rationale and design of a cluster-randomized multifaceted intervention trial to improve stroke care quality in China: The GOLDEN BRIDGE-Acute Ischemic Stroke. Am Heart J. 2015 Jun;169(6):767-774.e2. doi: 10.1016/j.ahj.2015.03.008. Epub 2015 Mar 26. PMID 26027613
- [Background] Wardlaw JM, Brazzelli M, Chappell FM, Miranda H, Shuler K, Sandercock PA, Dennis MS. ABCD2 score and secondary stroke prevention: meta-analysis and effect per 1,000 patients triaged. Neurology. 2015 Jul 28;85(4):373-80. doi: 10.1212/WNL.0000000000001780. Epub 2015 Jul 1. PMID 26136519
- [Background] Song B, Fang H, Zhao L, Gao Y, Tan S, Lu J, Sun S, Chandra A, Wang R, Xu Y. Validation of the ABCD3-I score to predict stroke risk after transient ischemic attack. Stroke. 2013 May;44(5):1244-8. doi: 10.1161/STROKEAHA.113.000969. Epub 2013 Mar 26. PMID 23532014
- [Background] Wang Y, Zhao X, Liu L, Soo YO, Pu Y, Pan Y, Wang Y, Zou X, Leung TW, Cai Y, Bai Q, Wu Y, Wang C, Pan X, Luo B, Wong KS; CICAS Study Group. Prevalence and outcomes of symptomatic intracranial large artery stenoses and occlusions in China: the Chinese Intracranial Atherosclerosis (CICAS) Study. Stroke. 2014 Mar;45(3):663-9. doi: 10.1161/STROKEAHA.113.003508. Epub 2014 Jan 30. PMID 24481975
- [Background] Suri MF, Qiao Y, Ma X, Guallar E, Zhou J, Zhang Y, Liu L, Chu H, Qureshi AI, Alonso A, Folsom AR, Wasserman BA. Prevalence of Intracranial Atherosclerotic Stenosis Using High-Resolution Magnetic Resonance Angiography in the General Population: The Atherosclerosis Risk in Communities Study. Stroke. 2016 May;47(5):1187-93. doi: 10.1161/STROKEAHA.115.011292. Epub 2016 Apr 7. PMID 27056984
- [Background] Amarenco P, Lavallee PC, Labreuche J, Albers GW, Bornstein NM, Canhao P, Caplan LR, Donnan GA, Ferro JM, Hennerici MG, Molina C, Rothwell PM, Sissani L, Skoloudik D, Steg PG, Touboul PJ, Uchiyama S, Vicaut E, Wong LK; TIAregistry.org Investigators. One-Year Risk of Stroke after Transient Ischemic Attack or Minor Stroke. N Engl J Med. 2016 Apr 21;374(16):1533-42. doi: 10.1056/NEJMoa1412981. PMID 27096581
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Wang Y, Pan Y, Zhao X, Li H, Wang D, Johnston SC, Liu L, Meng X, Wang A, Wang C, Wang Y; CHANCE Investigators. Clopidogrel With Aspirin in Acute Minor Stroke or Transient Ischemic Attack (CHANCE) Trial: One-Year Outcomes. Circulation. 2015 Jul 7;132(1):40-6. doi: 10.1161/CIRCULATIONAHA.114.014791. Epub 2015 May 8. PMID 25957224